CLINICAL TRIAL: NCT02164409
Title: Next-Generation Sequencing to Evaluate Transcriptomic Changes Associated With H. Pylori Infection and Gastric Cancer Carcinogenesis
Brief Title: Changes Associated With H. Pylori and Gastric Carcinogenesis
Acronym: IIT H pylori
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1203012274
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To examine RNA tranome of gastric cancer mucosa, in patients with H. pylori infection & examine spectrum of disease associated with infection. We will also examine bacterial content of samples to pinpoint specific H. pylori strain(s) & stomach microbial profile to correlate with gastric mucosal tranome & predisposition of gastric cancer. We plan to take 2-3 additional biopsies from an area of stomach already being sampled. The biopsies will be used for next-generation RNA & DNA sequencing & novel bioinformatics analyses. Examination of the genetic impact of H. pylori infection in patients may expose genetic factors that influence gastric cancer carcinogenesis & give deeper insight into molecular pathways that serve as candidate biomarkers for gastric cancer carcinogenesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Subjects for this study will be either H. pylori positive with an active infection, cleared of an H. pylori infection or be both H. pylori antibody positive and have a malignancy of the gastrointestinal tract, specifically gastric adenocarcinoma.
  Interventions: Procedure: Endoscopy tissue collection
- Control: A small subset of patients without H. pylori infection will be enrolled as well (n=30) to serve as a control group.
  Interventions: Procedure: Endoscopy tissue collection

INTERVENTIONS:
Procedure: Endoscopy tissue collection — The investigational part of this study is the requirement for an additional biopsy from a site that is already being biopsied at the time of a routine endoscopy. Any patients who develop bleeding following their routine clinical biopsies will not undergo any additional research biopsies.

SUMMARY:
This is a research study for patients who currently have or previously had an H. pylori infection or who have gastric or esophageal cancer and who plan to undergo an endoscopy as part of their care. The purpose of this study is to find out how and why H. pylori infections can cause progression to gastric cancer and if it's possible for intervention prior to this progression.

DETAILED DESCRIPTION:
H. pylori infection is a prevalent environmental cause of gastric cancer. The molecular mechanisms of carcinogenesis due to H. pylori remain unexplained and consequences of infection are variable and unpredictable. The aim of this research is to examine the RNA transcriptome of gastric cancer mucosa (gastric mucosa is the mucus membrane of the stomach), in patients with H. pylori infection and examine the spectrum of disease associated with infection. We will also examine bacterial content of samples to pinpoint the specific H. pylori strain(s) and the stomach microbial profile to correlate with the gastric mucosal transcriptome and predisposition of gastric cancer. Patients with prior or current active H. pylori infection who are planning to under endoscopic evaluation will be eligible for participation. From these patients, we plan to take up to four additional biopsies from each area of stomach already being sampled.

The biopsies will be used for next-generation RNA and DNA sequencing and novel bioinformatics analyses. The analysis will be performed at Weill Cornell Medical College by Doron Betel, PhD. The sequencing will be performed in the Epigenetics Core laboratory under the supervision of Doron Betel, who will be working closely with the principal investigator, Manish A. Shah, M.D. Examination of the genetic impact of H. pylori infection in patients may expose genetic factors that influence gastric cancer carcinogenesis and give deeper insight into molecular pathways that serve as candidate biomarkers for gastric cancer carcinogenesis. Our goal is to distinguish patients with chronic H. pylori infection who are at risk of subsequently developing gastric cancer from the vast majority of patients with H. pylori infection who do not develop malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years or older
* Patient must have active or prior H. pylori infection, or have been treated for H.pylori infection in the past, as assessed by ELISA (not applicable for the subset of patient controls) or have gastric or esophageal cancer or have Barrett's Esophagus
* Patients must be eligible for and are planning to undergo a routine upper endoscopy and tissue biopsy
* Patients must sign informed consent

Exclusion Criteria:

* Prior history of upper GI bleed (within 3 months)
* Bleeding disorder or coagulopathy
* Recent stroke or myocardial infarction (within 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will be either H. pylori positive with an active infection, cleared of an H. pylori infection or be both H. pylori antibody positive and have a malignancy of the gastrointestinal tract, specifically gastric adenocarcinoma. Of note, a small subset of patients without H. pylori infection will be enrolled as well (n=30) to serve as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Identify genomic alterations associated with H. pylori infection | Within 3 years of tissue collection
  Ability to obtain adequate tissue for next generation sequencing from endoscopy

SECONDARY OUTCOMES:
Examine bacterial content in samples | at time of sample collection
  High-throughput DNA and RNA sequencing will be used to determine bacterial content of samples

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No